CLINICAL TRIAL: NCT06443411
Title: R&D of Non-invasive Innovative Intracranial Waves Monitoring System for Diagnostics and Treatment Monitoring of Patients with Normal Tension Glaucoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Kaunas University of Technology (Other)
Responsible Party: Principal Investigator, Ugne Kevalaite, Medical Doctor, Lithuanian University of Health Sciences
Other Study IDs: 2024-BE10-0001
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-05

CONDITIONS: Normal Tension Glaucoma
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Glaucoma group: The prospective clinical study will include at least 56 patients with NTG using non-invasive ICP waves monitoring system through a human eye orbit without applying external pressure to the eye with approximately 10 millisecond temporal resolution. It is a prospective longitudinal study of patients with normal tension glaucoma by the inclusion age from 25 to 65 years. The standard monitoring session will last 1-3 minutes. Sex: male and female. Exclusion criterion is documented neurodegenerative disorders.
  Interventions: Other: Monitoring of cerebral hemodynamics
- Control group: 100 healthy subjects using non-invasive ICP waves monitoring system through a human eye orbit without applying external pressure to the eye with approximately 10 millisecond temporal resolution.
  Interventions: Other: Monitoring of cerebral hemodynamics

INTERVENTIONS:
Other: Monitoring of cerebral hemodynamics — A specially designed pair of goggles will be put on the patient's head. The closed eyelids, along with the surrounding tissues, will be in contact with a thin, elastic, non-allergic film used to seal water filled inside the goggles. Pulse waves, including those originating from cerebrospinal fluid pulsation, will be transmitted from the eyelids to the water, where they will be detected by a pressure sensor and recorded with a laptop.

SUMMARY:
Assessment and monitoring of intracranial pressure (ICP) changes are important in the management of cerebral pathologies. In the eye, ICP increase and decrease both correlate with optic neuropathies, the former because of papilledema and the latter related to glaucoma. While the relationship between ICP elevation and papilledema is well established, the relationship between low ICP and glaucoma is still poorly understood. So far, ICP monitoring is performed invasively, but this entails risks including infection, spurring the study of non-invasive alternatives. While none of currently methods in use can fully replace invasive techniques, certain measures show great potential for specific applications. In this context, monitoring the intracranial pressure changes of normal tension glaucoma may lead to a better understanding of how intracranial pressure waves vary in normal tension glaucoma. Treatment of normal tension glaucoma as a two-pressure disease needs periodic intracranial dynamic monitoring sessions for evaluation of treatment effectiveness and for needed corrections of treatment methodology.

Project aim is to be able to monitor the "missing link" of intracranial dynamics of patients with normal tension glaucoma according to circadian rhythm: in the morning, during lunch and in the evening. The opportunity to monitor ICP waves non-invasively for patients with normal tension glaucoma will be implemented for the first time by using novel non-invasive intracranial pressure waves real-time monitoring system invented by KTU team in 2022 (patent applications are in the process of registration in the EU and USA).

ELIGIBILITY:
Inclusion Criteria:

* 25-65 years of age.
* The patient, after reading the personal information form, confirms in writing his / her consent to participate in the study.
* The study group includes patients with a primary open-angle normal intraocular pressure glaucoma diagnosis confirmed by an ophthalmologist (typical glaucomatous changes in the optic nerve disc and eye area, open angle of the anterior chamber, intraocular pressure in the diurnal curve with/without anti-glaucoma medication ≤ 21 mmHg) and IOP ≤ 21mmHg on study day with/without anti-glaucoma medication.
* The control group includes healthy volunteers who do not suffer from glaucoma, acute or chronic uncompensated disease that may affect the results of the research, and according to age and anthropometric data correspond to the individuals of other research groups.

Exclusion Criteria:

* Patient's refusal to participate in biomedical research.
* Persons younger than 25 years or older than 65 years.
* A woman who may become pregnant, be pregnant or breastfeeding.
* The patient is allergic or sensitive to local anesthetics.
* Suffering from an eye disease that may distort the results of the study, if so decided by the examining physician.
* Patients who have had orbital or eye trauma.
* Patients who have undergone any eye surgery.
* Patients with acute or chronic, but currently aggravated, respiratory system disease.
* Patients with uncompensated cardiovascular diseases (II-III AV block or cardiogenic shock).
* Patients with uncompensated diabetes.
* Neurological diseases, mental illnesses identified in the anamnesis.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients treated at the Clinic of Eye Diseases, Hospital of Lithuanian UHS.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-12-22 (Estimated); Study Completion 2025-02-22 (Estimated)

PRIMARY OUTCOMES:
A validated non-invasive ICP waves real-time monitoring technology | From 2024-04-22 till 2025-02-22
  Validation of non-invasive ICP waves real-time monitoring through a human eye orbit without applying external pressure to diagnose NTG with the required sensitivity and specificity to make treatment decisions.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania